CLINICAL TRIAL: NCT07343349
Title: Addition of Focal Boost to Primary Radiotherapy for Prostate Cancer in 12 or 20 Fractions: A Large DAPROCA Randomised Trial.
Brief Title: Addition of Focal Boost to Primary Radiotherapy for Prostate Cancer in 12 or 20 Fractions
Acronym: DAPROCA10
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Sygehus Lillebaelt (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Copenhagen University Hospital at Herlev (Other); Naestved Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Peter Meidahl Petersen, MD, Ph.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-25028267
Record Dates: First submitted 2025-12-02; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Patients Undergoing External Radiation and Seed Implantation; High Risk Localised Prostate Carcinoma; Locally Advanced Prostate Cancer; Unfavourable Intermediate Risk Prostate Cancer
Keywords: Prostate cancer; Radiotherapy; Hypofractionation; Boost
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial is an open, randomised, 2 x 2 factorial design, randomising between:
  1. Boost or no boost to intra-prostatic tumour lesions.
  2. 20 fractions in 4 weeks versus 12 fractions in 2½ weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 20 treatment fractions no boost (Active Comparator): Prostate and seminal vesicles: 60 Gy/ 20 fractions. Pelvic: 45 Gy /20 fractions.
  Interventions: Radiation: Addition of focal boost and hypofractionation
- 20 treatment fractions, boost (Experimental): Boost to intra-prostatic lesions: 75 Gy/20 fractions, prostate and seminal vesicles: 60 Gy/ 20 fractions. Pelvic: 45 Gy /20 fractions.
  Interventions: Radiation: Addition of focal boost and hypofractionation
- 12 treatment fractions, no boost (Experimental): Prostate and seminal vesicles: 50 Gy/ 12 fractions, Pelvic: 37 Gy /12 fractions.
  Interventions: Radiation: Addition of focal boost and hypofractionation
- 12 fractions, boost (Experimental): Boost to intraprostatic lesions: 60 Gy/12 fractions, prostate and seminal vesicles: 50 Gy/12 fractions, pelvic: 37 Gy /12 fractions.
  Interventions: Radiation: Addition of focal boost and hypofractionation

INTERVENTIONS:
Radiation: Addition of focal boost and hypofractionation — Addition of focal boost to primary radiotherapy for prostate cancer in 12 or 20 fractions

SUMMARY:
Every year, about 700 Danish men get radiotherapy for prostate cancer with a high-risk of later progression. The risk of relapse is about 40 % after 5 - 8 years, so we need better treatment for these patients in Denmark and globally. The aim is to reduce later cancer spreading, need of hormone treatments and prostate cancer death.

DAPROCA 10 tests two possible improvements:

If a higher dose (boost) to intra-prostatic tumor lesions improves cure rates. If the radiotherapy can be given with 12 treatment fractions instead of 20 without increased side-effects.

In this randomised trial half the participants get a boost and the other half don't. Half the patients get 12 treatments, the other half 20.

To answer these questions we must include1016 participants. The trial is feasible because the technological advances in imaging and radiotherapy enables us to define the tumors in the prostate and to deliver the boost to the tumors with high precision, without increased dose to the surrounding organs.

DETAILED DESCRIPTION:
Addition of focal boost to primary radiotherapy for prostate cancer in 12 or 20 fractions: A large DAPROCA randomised trial.

Purpose

The DAPROCA multidisciplinary group is planning a large trial to answer two pertinent questions of how to improve radiotherapy for high - and intermediate risk prostate cancer:

1. Will increasing dose to intra-prostatic cancer lesions improve outcomes with respect to prostate cancer without increasing toxicity?
2. Is it possible to shorten the treatment without increased toxicity?

The success of both increased dose to intra-prostatic cancer lesions and shortening of treatment, which means treatment with fewer treatment fractions with higher dose per fraction, is most likely dependent on high quality, high precision radiotherapy (RT) planning and delivery. A French randomised trial in prostate cancer demonstrated improved rectal toxicity scores (p=<0.03) and biochemical control with image guidance, and the MIRAGE randomised trial demonstrated improvements with smaller margins and more precise delivery (1-3). Many European clinics, including the Danish RT-clinics are able to provide high quality RT to all patients as per national consensus guidelines and in this study, we aim to further develop and implement this high quality opportunities in order to deliver hypofractionated RT and to boost the dose to intraprostatic lesions in all participating centers.

Background Prostate cancer (PCa) is the second most common malignancy in men worldwide, and the most common cancer in Denmark. The incidence of PCa has been increasing in most coun-tries and varies between countries. In Denmark, the incidence is now 124/100.000 men per year, and the median age for men diagnosed with PCa is 72 years. In the public, PCa is con-sidered to have a good prognosis, but the fact is that the mortality is high with 1323 Danish men annually dying from PCa, exceeding the age-standardised breast cancer mortality (nordcan,https://nordcan.iarc.fr/en). The prognosis and the treatment of PCa depends on pa-tient factors, as well as the histology grade, the prostate specific antigen (PSA) level, and the extent of disease.

This trial focuses on the group of patients with intermediate and high risk PCa, who have a risk of relapse of 25 - 60% and a risk of getting metastatic disease of up to 20 % after 5 - 8 years.

Large, randomised trials have shown improved oncological outcomes, including overall sur-vival, and disease specific survival for RT combined with androgen deprivation therapy (ADT) compared to ADT only. In addition, large, randomised trials have shown a benefit with RT and ADT compared to RT only. In 2023 in Denmark, 463 high risk patients and 144 intermediate risk patients received definitive RT with 36+ fractions. The RT is delivered with intensity mod-ulated RT (IMRT) and with prostate implanted fiducial markers for image guidance (IGRT). The RT clinics follow national guidelines securing the quality of treatment.

Endocrine treatment Endocrine treatment in combination with definitive RT has been standard of care for many years. The addition of 6-36 months of ADT has been shown to significantly improve overall survival (OS) in high risk and selected intermediate risk patients. Recent results revealed that two years of abiraterone acetate plus 3 years of ADT further improved the OS in patients with lymph node involvement or in high risk patients patients with two of three risk factors (>=cT3a, PSA ≧ 40, ISUP>=4).

Elective pelvic lymph node radiotherapy Elective pelvic lymph node radiotherapy (PLNRT) is offered in Denmark as a standard of care to PCa patients referred to definitive RT with either pelvic lymph node metastases or patients with a risk of lymph node metastases above 5- 7%. Risk of lymph node metastases can be estimated using different nomograms e.g. the Roach Formula, the Briganti nomogram 2012, Briganti nomogram 2019, and the Briganti nomogram 2023. Risk estimation can be based on imaging with PSMA PET/CT, mpMRI, PSA level, ISUP grade, T stage, tumour size, and the percentage of systematic prostate core biopsies with cancer. The benefit of elective pelvic lymph node irradiation is dependent on the risk of lymph node involvement, the higher the risk of lymph node involvement the more likely the patient is to benefit. Trials indicate im-provement of outcome and pelvic nodes can be included safely with contemporary radiother-apy techniques with tolerable risks of gastro-intestinal toxicity and edema.

Increased dose to intra-prostatic cancer lesions A strategy to improve outcome is dose escalation to the cancer lesions in the prostate. The FLAME randomised trial (NCT01168479) demonstrated improved biochemical control, re-duced local failure (LF) and reduced regional + distant metastatic failure. Toxicity is the limit-ing factor, and the boost dose was strictly limited depending on organ at risk exposure (OAR) in the FLAME trial. A dose response analysis for biochemical control indicated that patients with higher achieved boost doses experienced better tumour control. At the same time, the data suggested reduced toxicity as a result of further consideration of radiation dose to OARs and improved urethral sparing in particular. The question is therefore whether the addition of a focal boost can be established as standard of care.

A study larger than FLAME is needed in order to confirm effectiveness with freedom from distant metastases (FFDM) as an improved primary endpoint, compared to biochemical con-trol which was used as primary endpoint in FLAME. However, while endpoints based on bio-chemical relapse free survival are not surrogate for overall survival in localised prostate can-cer, FFDM is now shown to be a valid surrogate endpoint for OS in trials of localised prostate cancer. Biochemical control is used as a secondary endpoint in the current study to confirm the FLAME results and study heterogeneity of treatment effects as detailed in the statistics section.

Shortening of treatment duration In recent years, different approaches have been taken to decrease the number of fractions of prostate RT. These schedules reduce the number of hospital visits for patient convenience and cost-efficiency improvements. The large randomised CHHiP trial has shown good results with a 20-fraction schedule, albeit excluding the very high-risk patients. One study compared 78 Gy in 39 fractions with 60 Gy in 20 fractions and shortening treatment was not inferior re-garding biochemical disease-free survival or toxicity. One phase III study in locally advanced disease showed more acute, but similar long-term gastro-intestinal toxicity with the same tu-mour control in patients treated with 64.6 Gy / 19 fractions than with 78 Gy/39 fractions. Early results of a high-risk patient only trial including 329 patients were published in May 2023, showing that moderate hypo-fractionation RT is well-tolerated, similar to standard fractiona-tion RT at 2 years. These findings are in agreement with a large meta-analysis concerning moderate hypofractionation for high-risk PCa patients who also received pelvic lymph node irradiation, with the conclusion that moderate hypofractionation could be considered an alter-native to standard fractionated RT.

Ultra-hypofractionation trials show promising results but are currently not conclusive enough to be considered standard of care. The second research question is therefore to ultimately investigate if a shorter treatment of patients with intermediate and high-risk PCa, including treatment to pelvic lymph nodes, can be introduced.

In our study, the dose to elective lymph nodes is either 45 Gy in 20 fractions (2.25 Gy per fraction) or 37 Gy in 12 fractions (3.08 Gy per fraction). The table below provides an over-view of selected studies in which fractionations between 2 - 5 Gy have been used for pelvic lymph node radiotherapy.

Imaging During the recent two decades, imaging procedures have shown to improve accuracy of staging in prostate cancer. T stage is still strictly based on digital rectal examination, however multiparametric MRI is now standard staging procedure in order to predict extra prostatic ex-tension, seminal vesicle involvement, T-staging and to guide biopsies. Recently, PET using radioactive ligands binding to the prostate-specific membrane antigen (PSMA) combined with CT (PSMA-PET/CT) has shown higher accuracy for N and M staging and PSMA-PET/CT is now according to international guidelines the recommended staging procedure N and M stage even though the prognosis and ideal management of patients diagnosed as metastatic by these more sensitive tests is unknown.

MRI has been shown to improve accuracy of prostate delineation and to correlate with histol-ogy and definition of intra-prostatic lesions with MRI has shown a high accuracy. Recently, the combination of PSMA-PET and MRI has demonstrated even higher accuracy.

Based on the randomised trials showing benefit of radiotherapy with combined hormone- and radiotherapy compared to hormone therapy only, 3 months pre-irradiation castration is stand-ard for high-risk patients in many institutions. Studies have addressed weakening MRI signals and PSMA PET-uptake after castration. However, there is not enough data to guide us to the optimal imaging to define intra-prostatic lesions in patients who are treated with a combination of medical castration and radiotherapy. Currently this topic is being investigated in a phase 2 study (Danish Ethical Committee 2303938), conducted by the research group to prepare for the present study.

Additional improvements in delivery, such as MRI based image guidance, improved CT based image guidance, or adaption of the daily dose plan to the anatomy of the day etc. may improve outcomes further. If participating centers implement follow local adaptive strategies for adaptation due to anatomical changes, the center must document the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy verified PCa with no distant metastases with either
* Intermediate- or high-risk PCa, defined as at least one of the following risk criteria:

  * Clinical stage cT2c-T3b (UICC TNM 8th edition)
  * Imaging stage, T3a or T3b
  * ≥ Gleason score 4+3, (ISUP Grade groups 3,4 or 5)
  * Regional lymph node metastases N1
* Age > 18
* WHO score 0-1
* Intraprostatic lesion visible on MRI
* Suitable for focal boost
* Ability to give written informed consent and willingness to return for follow-up

Exclusion Criteria:

* WHO performance status ≥ 2
* If, for any patient related reason, an MRI cannot be performed
* T4
* International prostate symptom score (IPSS) ≧ 20
* If fiducial markers cannot be inserted
* TURP within 3 months from start of treatment
* Previous pelvic irradiation
* If the patient is judged by the physician to be unable to adhere to trial activities
* History of chronic inflammatory bowel disease (CIBD)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2040-10-30 (Estimated); Study Completion 2040-10-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from distant metastasis | Time from enrollment to confirmation of occurence of radigraphic distant metastases. The patients are followed for 123 months after start of radiotherapy.
  Metastses is verified by PSMA scan which is recommended:
  * If a recurrence is suspected biochemically according to biochemical relaps accordingly to the Phoenix criteria
  * If a recurrence is suspected clinically, e.g: Bone pain, anemia, urinary symptoms
  * If recurrence is suspected by radiographic test Biopsy is also accepted and MRI, CT, bone scintigraphy, NAF-PET, ultrasound or clinical examination may also be accepted with further confirmation, e.g. biopsy or laboratory tests.
  If the event "distant metastasis" is based on tests without biopsy or PSMA positivity the event shall be confirmed at a multi-disciplinary tumor board.

SECONDARY OUTCOMES:
Freedom from biochemical relapse | Time from enrollment to confirmation of occurence of biochemical relapse. PSA is measured by a blood test regularly until 123 months after start of radiotherapy.
  Phoenix criteria are used for definition of the event biochemical relapse, defined as a PSA increase of 2 ug/l from nadir. The date of recurrence is the first date with a PSA level of nadir + 2. The PSA level must be confirmed by a second PSA measurement performed at minimum two weeks later.
Time to salvage hormonal therapy | Time from enrollment to intiation of salvage hormonal therapy. Hormone treatment is recordet at regular patient visits until 123 months after start of radiotherapy.
  Any hormone treatment will be recorded at follow-up visits and date will be verifed by the date of treatment start in the eletronic medicins system.
Regional relapse-free survival | Time from enrollment to confirmation of regional relapse-free survival. Time Frame: The patients are followed for 123 months after start of radiotherapy.
  Regional metastses means recurrence in lymph nodes is verified by PSMA scan which is recommended:
  * If a recurrence is suspected biochemically according to the Phoenix criteria
  * If a recurrence is suspected clinically, e.g: Bone pain, anemia, urinary symp-toms
  * If recurrence is suspected by radiographic test Biopsy is also accepted and MRI, CT, ultrasound or clinical examination may also be accepted with further confirmation, e.g. biopsy or laboratory tests.
  If the event "regional metastasis" is based on tests without biopsy or PSMA positivity the event shall be confirmed at a multi-disciplinary tumor board.
Local relapse-free survival | Time from enrollment to confirmation of local relapse. The participants are followed for 123 months after start of radiotherapy
  The event local recurrence is defined as a local PSMA positive lesion. Local recurrence after definitive radiotherapy should be confirmed by biopsy from the site of suspected recurrence. MRI, CT, ultrasound or clinical examination may also be accepted with further confirmation, e.g. biopsy.
Overall survival | Time from enrollment to death of any cause. Cause and time of death is collected for up to 20 years.
  Cause and time of death is collected from electronic patient charts. If no information is available, data will be retrieved from the national death register.
Prostate cancer specific survival | Time from enrollment to death of prostate cancer. Cause and time of death is collected for up to 20 years.
  Time of death from prostate cancer is collected from electronic patient charts. If no information is available, data will be retrieved from the national death register.
Self-reported quality of life | Reported at baseline and 3 months, 1 year, 2 years 5 years after start of radiotherapy.
  Using the tested and validated EORTC QLQ-PR25 questionnaire.
Self reported quality of life | Reported at baseline and 3 months, 1 year, 2 years 5 years after start of radiotherapy.
  Using the tested and validated EORTC QLQ-C30 questionnaire.
Toxicity as CTCAE | Reported at baseline and 3 months, 1 year, 2 years 5 years after start of radiotherapy.
  CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aurhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sygehus Lillebaelt, Vejle

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted in accordance with European General Data Protection Regulation. We intend to share data in anonymous form.
  The statistical analysis plan is described in the attached study protocol.
Supporting Information: Study Protocol
Time Frame: Not decided yet.
Access Criteria: Not decided yet.

DOCUMENTS (1):
  • Study Protocol (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT07343349/Prot_000.pdf